CLINICAL TRIAL: NCT03171857
Title: Role of Doppler Ultrasound in Evaluation of Superficial Soft Tissue Masses
Brief Title: Doppler Ultrasound in Characterization of Superficial Soft Tissue Masses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Samir, principal investigator, Assiut University
Other Study IDs: DUSSSTM
Record Dates: First submitted 2017-05-28; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Mass of Soft Tissue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A wide variety of superficial soft tissue masses may be seen in clinical practice. Superficial soft tissue masses can generally be categorized as mesenchymal tumors, skin appendage lesions, metastatic tumors, other tumors and tumor-like lesions, or inflammatory lesions. The investigators will use doppler ultrasound in evaluation of superficial soft tissue masses characterization.

DETAILED DESCRIPTION:
There are many examples for these benign superficial soft tissue lesions as lipoma, ganglion, Baker's cyst, giant cell tumor, lymphangioma, hernia, abscess, epidermoid cyst, hematoma, muscle rupture, glomus tumor, fibromatosis, lymphadenitis hemangioma, exostosis, fibroma, neurofibroma and schwannoma. Malignant lesions also could be seen as lymphoma, metastasis, osteogenic sarcoma, liposarcoma , leiomyosarcoma, rhabdomyosarcoma and synovial sarcoma.

Nowadays, High resolution ultrasound has a high sensitivity in detecting superficial soft tissue masses through the grey-scale grading that compose an image range from pure black at the weakest intensity to pure white at the strongest that can be used to evaluate its structure, some aspects of its function and to determine the nature of a mass lesion (cystic or solid) and with Doppler ultrasound which is an excellent imaging modality to determine the vascularity of superficial soft tissue masses that can be characterized in terms of their echogenicity, margin, shape, composition, acoustic transmission, size, the grading of color Doppler ultrasound , and resistive index in spectral Doppler as spectral Doppler will be applied in lesions with positive color flow signals.

ELIGIBILITY:
Inclusion Criteria:

* Patients in different age groups with superficial soft tissue lesions

Exclusion Criteria:

* If the patient undergo previous operations at the same mass that could change the criteria of that mass or if the mass is recurrent at the same site.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that have superficial soft tissue masses in different age groups that referred from the outpatient clinics of the general or orthopaedic surgery, Assiut University Hospital to the Diagnostic Radiology Department
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Patients diagnosed as superficial soft tissue lesions by doppler ultrasound. | 2 years
  Effectiveness of Doppler ultrasound in evaluation of superficial soft tissue masses in comparison with histopathological data of these lesions.

REFERENCES:
- [Background] Brkljacic B, Kuzmic AC, Dmitrovic R, Rados M, Vidjak V. Doppler sonographic renal resistance index and resistance index ratio in children and adolescents with unilateral hydronephrosis. Eur Radiol. 2002 Nov;12(11):2747-51. doi: 10.1007/s00330-001-1259-0. Epub 2002 Feb 2. PMID 12386768
- [Background] Taurino M, Rizzo L, Stella N, Mastroddi M, Conteduca F, Maggiore C, Faraglia V. Doppler ultrasonography and exercise testing in diagnosing a popliteal artery adventitial cyst. Cardiovasc Ultrasound. 2009 May 27;7:23. doi: 10.1186/1476-7120-7-23. PMID 19473494
- [Background] Toprak H, Kilic E, Serter A, Kocakoc E, Ozgocmen S. Doppler US in rheumatic diseases with special emphasis on rheumatoid arthritis and spondyloarthritis. Diagn Interv Radiol. 2014 Jan-Feb;20(1):72-7. doi: 10.5152/dir.2013.13127. PMID 23996840